CLINICAL TRIAL: NCT05955196
Title: Test of CD47-SIRPα Inhibitors on the Immune Microenvironment Colon Cancer
Acronym: MACROSWITCH
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: MACROSWITCH-IPC 2021-083
Record Dates: First submitted 2023-01-27; First posted 2023-07-21 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Cancer of the Colon
MeSH Terms: conditions — Colonic Neoplasms | interventions — Tumor Burden

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — peripheral blood; samples of colon cancers with healthy tissue in parallel on the surgical specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: BLOOD AND TUMOR — sampling of 24 ml of peripheral blood and samples of colon cancers with healthy tissue in parallel on the surgery piece

SUMMARY:
Our goal is to create novel CD47-SIRPα inhibitors using small molecules to reverse TAM-mediated immune suppression and restore anti-tumor immunity in CRCs. Our program uses structure-based drug design to create selective and potent small molecule inhibitors of SIRPα-CD47 to target the tumor microenvironment with greater efficacy and lower toxicity than CD47-targeting antibodies. .

In order to study the activity of CD47-SIRPα inhibitors on the immune microenvironment of tumors, we propose to use organoids derived from biopsies of patients with colon cancer. Tumoroids preserve the patient's tumor stroma (including myeloid cells) and provide an accurate in vitro model of complex tumor immune interaction for the evaluation of immunotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient who has signed a consent to participate;
* Patient with metastatic or non-metastatic colon cancer, or recurrence of colon cancer for whom excision surgery has been proposed;
* Patient affiliated to a social security scheme, or beneficiary of such a scheme

Exclusion Criteria:

* Patient who had emergency colon cancer surgery
* Person in an emergency situation or unable to express their consent.
* Adult subject to a legal protection measure (adult under guardianship, curatorship or safeguard of justice),
* Patient unable to submit to the medical follow-up of the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied concerns patients over the age of 18, suffering from colon cancer, undergoing immediate surgery or after chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-01-09 (Estimated); Study Completion 2027-01-09 (Estimated)

PRIMARY OUTCOMES:
Establishment of patient derived organoids (minimum n=30) resembling the primary tissue sample | 18 months from study launch
  the capacity to establish patient-derived organoids from tumor and adjacent normal tissue will be evaluated using a histology score evaluating and comparing primary and organoid sample characteristics.

SECONDARY OUTCOMES:
Establishment of a validated cryobank of patient derived organoids (minimum n=30) | 18 months from study launch
  the capacity to establish a cryobank of patient-derived organoids from tumor and adjacent normal tissue will be evaluated using a growth score evaluating and comparing organoid sample characteristics pre- and post-cryopreservation and amplification through 4 passages.
Generate a T cell biobank by FACS isolating T cells using the CD3 surface marker directed against the human form | 48 month
To assess the effect of immunotherapy on the antitumor activity of autologous T cells from peripheral blood samples using tumor viability measurements (cell titer glo, FACS) | 48 month

CONTACTS AND LOCATIONS:
Overall Officials: Cécile de CHAISEMARTIN, MD, Principal Investigator — Paoli Calmettes Institute
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No